CLINICAL TRIAL: NCT02869984
Title: Clinical Trial Assessing 5-HT3 Receptor Antagonist (Ramosetron) for the Treatment of Anterior Resection Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A ST (Unknown)
Responsible Party: Principal Investigator, Kyu Joo Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1604-095-755
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Anterior Resection Syndrome
MeSH Terms: interventions — ramosetron

ARMS (2):
- Treatment (Experimental): ramosetron treatment for 4 weeks from 1mo after anterior resection for rectal cancer
  Interventions: Drug: Ramosetron
- Control (No Intervention): No treatment

INTERVENTIONS:
Drug: Ramosetron
  Arms: Treatment

SUMMARY:
Poor functional outcomes has been reported inevitably, and up to 90% of the patients have experienced bowel habit changes after sphincter-saving surgery for rectal cancer. But, currently there has been no specific treatment for ARS and symptom based empirical management is tried Recently, 5-HT3 receptor antagonists can be used for treatment of IBS-D, and has been revealed to be slowing the bowel movement and improving stool consistency and urgency.

We performed the clinical trial with using ramosetron (Irribow®) for the treatment of ARS

ELIGIBILITY:
Inclusion Criteria:

* The patients who undergo sphincter saving surgery for rectal cancer

Exclusion Criteria:

* recurred rectal cancer
* rectal cancer with distant metastasis
* permanent stoma formation
* postoperative concurrent chemoradiotherapy
* uncontrolled medical disease
* inflammatory bowel disease
* uncontrolled constipation
* preoperative incontinence (LARS score, more than 20)
* allergic to intervention drug

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
low anterior resection syndrome score | 4 weeks
  questionnaire with comparison of frequency or urgency

SECONDARY OUTCOMES:
Quality of Life score | 4 weeks
  EORTC QLQ C30 (Korean version, validated)

REFERENCES:
- [Derived] Ryoo SB, Park JW, Lee DW, Lee MA, Kwon YH, Kim MJ, Moon SH, Jeong SY, Park KJ. Anterior resection syndrome: a randomized clinical trial of a 5-HT3 receptor antagonist (ramosetron) in male patients with rectal cancer. Br J Surg. 2021 Jun 22;108(6):644-651. doi: 10.1093/bjs/znab071. PMID 33982068